CLINICAL TRIAL: NCT06844708
Title: CMTS0929 for Inflammatory Bowel Disease: a Prospective, Open-label, Single-arm Clinical Study
Brief Title: CMTS0929 for Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024CMTS0929-IBD
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: inflammatory bowel disease; CMTS0929; efficacy; safety
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive treatment with CMTS0929. They will be administered one unit of the liquid via colonic transendoscopic enteral tube (cTET) for three consecutive days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Eligible subjects will receive treatment with China Microbiota Transplantation System 0929 (CMTS0929). They will be administered one unit of the liquid via colonic transendoscopic enteral tube (cTET) for three consecutive days.
  Interventions: Biological: CMTS0929

INTERVENTIONS:
Biological: CMTS0929 — China Microbiota Transplantation System 0929 (CMTS0929) is defined as suspension from washed microbiota.

SUMMARY:
This is a prospective, open-label, single-arm study to explore the safety and the efficacy of China Microbiota Transplantation System 0929 (CMTS0929) for patients with inflammatory bowel disease (IBD).

DETAILED DESCRIPTION:
At least 12 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. Data of demographic characteristics and clinical data will be collected. After treatment, they will enter the follow-up period for safety and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to enter the study:

1. Patients diagnosed with inflammatory bowel disease (IBD) based on typical clinical symptoms, endoscopic findings, and histological criteria.
2. Aged between 18 and 75 years old, regardless of gender.
3. No history of using antibiotics, prebiotics, or probiotics within at least the past month.
4. Patients who can fully understand the content of the informed consent form for this trial and voluntarily sign the written informed consent.
5. Patients willing to undergo subsequent follow - up and comply with other requirements of the protocol.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria must be excluded from the study:

1. Women who are pregnant or plan to become pregnant during the trial.
2. Patients who have any doubts about this technology or have a history of other risks.
3. Patients in the terminal stage of the disease or who may die during the study.
4. Patients with a history of antibiotic use within three months before transplantation or who have participated in other clinical trials.
5. Patients who have participated in any other microbiota - based therapies before enrollment.
6. Patients with positive antibodies for hepatitis B, tuberculosis, syphilis, or HIV, or those in the acute phase of any infectious disease.
7. Patients with cardiac function at grade III or higher, elevated transaminases more than twice the upper limit of the normal range, or renal insufficiency (glomerular filtration rate (GFR) less than 60 ml/min).
8. Patients with a fever of over 38 °C or clinically obvious active infections that may affect this trial.
9. Patients with severe anemia (hemoglobin < 60 g/L), granulocytopenia (absolute neutrophil count < 1.5×10⁹/L), or prolonged prothrombin time (PT) by more than 1.5 seconds.
10. Patients with obvious cardiovascular and cerebrovascular abnormalities (such as tachycardia or uncontrolled atrial fibrillation, acute coronary syndrome, stroke, or recurrent transient ischemic attacks (TIAs)); a history of arrhythmia (multifocal ventricular premature beats, bigeminy, trigeminy, congenital long QT syndrome), or patients with heart diseases that, in the judgment of the researcher, increase the risk of ventricular arrhythmia.
11. Situations identified by the researcher during the trial that may affect the patient's compliance and/or the completion of trial - related procedures, or clinical contraindications related to the pre - trial.
12. Patients who have undergone abdominal organ surgery within three months before treatment, patients less than 6 weeks after major organ surgery, or patients with poor wound healing after surgery.
13. Patients with gastrointestinal obstructive diseases, tumors, or hepatic or renal insufficiency.
14. Pregnant or lactating women, or women with the intention of becoming pregnant.
15. Patients suspected or confirmed to be drug users, or those with a history of immunodeficiency (such as positive HIV antibodies or currently receiving immunosuppressive therapy).
16. Patients with known major active infections, or those with major disorders in blood, renal, metabolic, gastrointestinal, or endocrine functions as judged by the researcher.
17. Other situations deemed unsuitable for enrollment by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy of China Microbiota Transplantation System 0929 (CMTS0929) | Four-week
  Partial Mayo scale for Ulcerative Colitis (UC), the minimum score is 0, the score ≤2 and no single sub-score was >1 is clinical remission, 3-5 as mild activity, 6-10 as moderate activity, 11-12 as severe activity.
The efficacy of China Microbiota Transplantation System 0929 (CMTS0929) | Four-week
  Crohn disease activity index (CDAI) for Crohn's disease (CD), the minimum value is 0, ≤ 4 is remission，5-7 is mild，8-16 is moderate, > 16 is severe, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The changes in endoscopic score | Three-month, Six-month
The change in hematochezia compared with baseline | One-week, Four-week, Twelve-week, Six-month
  Hematochezia can be evaluated by Fecal occult blood test (FOBT) and the record of gross blood stool. The frenquence of hematochezia should be recorded.
The change in frequency of defecation compared with baseline | One-week, Four-week, Twelve-week, Six-month
  The frequency of defecation per day should be recorded.
The change in abdominal pain compared with baseline | One-week, Four-week, Twelve-week, Six-month
  The abdominal pain should be recorded, such as 0 for none, 1 for mild, 2 for moderate, 3 for severe, 4 for very severe.
The incidence of IBD-related complications | One-week, Four-week, Twelve-week, Six-month
  Intestinal perforation, massive gastrointestinal bleeding, megacolon, malignancies associated with colorectal cancer or small intestine cancer
The rate of surgical intervention | Six-month
The safety of CMTS0929 | Immediately, One-week, Two-week, Four-week, Three-month, Six-month
  The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0: The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wortelboer K, de Jonge PA, Scheithauer TPM, Attaye I, Kemper EM, Nieuwdorp M, Herrema H. Phage-microbe dynamics after sterile faecal filtrate transplantation in individuals with metabolic syndrome: a double-blind, randomised, placebo-controlled clinical trial assessing efficacy and safety. Nat Commun. 2023 Sep 12;14(1):5600. doi: 10.1038/s41467-023-41329-z. PMID 37699894
- [Background] Shaukat A, Shyne M, Mandel JS, Snover D, Church TR. Colonoscopy With Polypectomy Reduces Long-Term Incidence of Colorectal Cancer in Both Men and Women: Extended Results From the Minnesota Colon Cancer Control Study. Gastroenterology. 2021 Mar;160(4):1397-1399.e3. doi: 10.1053/j.gastro.2020.11.014. Epub 2020 Nov 17. No abstract available. PMID 33217449
- [Background] Zhang F, Cui B, He X, Nie Y, Wu K, Fan D; FMT-standardization Study Group. Microbiota transplantation: concept, methodology and strategy for its modernization. Protein Cell. 2018 May;9(5):462-473. doi: 10.1007/s13238-018-0541-8. Epub 2018 Apr 24. PMID 29691757
- [Background] Piovani D, Hassan C, Repici A, Rimassa L, Carlo-Stella C, Nikolopoulos GK, Riboli E, Bonovas S. Risk of Cancer in Inflammatory Bowel Diseases: Umbrella Review and Reanalysis of Meta-analyses. Gastroenterology. 2022 Sep;163(3):671-684. doi: 10.1053/j.gastro.2022.05.038. Epub 2022 May 26. PMID 35643170
- [Background] Ungaro R, Mehandru S, Allen PB, Peyrin-Biroulet L, Colombel JF. Ulcerative colitis. Lancet. 2017 Apr 29;389(10080):1756-1770. doi: 10.1016/S0140-6736(16)32126-2. Epub 2016 Dec 1. PMID 27914657
- [Background] Hodson R. Inflammatory bowel disease. Nature. 2016 Dec 21;540(7634):S97. doi: 10.1038/540S97a. No abstract available. PMID 28002398